CLINICAL TRIAL: NCT06551272
Title: Microbiota Modification for Immuno-oncology in Hepatocellular Carcinoma
Acronym: MOTHER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Center Eugene Marquis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1-69-001
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: Immunotherapy; microbiome; resistance; dysbiosis; Faecalibacterium prausnitzii
MeSH Terms: conditions — Carcinoma, Hepatocellular; Dysbiosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- standard-of-care approved first-line immunotherapy- EXL01 (Experimental): Patients treated with atezolizumab-bevacizumab ou durvalumab with the addition of the experimental treatment exl01, 1 capsule per day for a maximum of 12 months.
  Interventions: Drug: EXL01

INTERVENTIONS:
Drug: EXL01 — EXL01 contains an unmodified single strain of F. prausnitzii

SUMMARY:
Hepatocellular carcinoma (HCC) is the most common liver primary cancer with a high rate of mortality. Since the results of IMbrave150, immunotherapy have emerged as a standard of care for HCC patients advanced and/or unresectable in first line of treatment. The objective response rate was about 30%, but half of patients would present only stable disease and about 20% progressive disease.

Faecalibacterium prausnitzii is one of the most abundant bacterial in human gut microbiota, around 5% of total bacteria in feces.

For patients with metastatic melanoma, treated with ipilimumab, an antibody targeting CTLA-4 (Cytotoxic T-lymphocyte-associated antigen 4), patients with a baseline gut microbiota enriched with Faecalibacterium had a significantly better clinical outcomes. In patients with metastatic melanoma, the level of Faecalibacterium prausnitzi at baseline was predictive of response to anti-PD-1 (programmed death-1) or anti-CTLA-4 therapy. EXL01 is a pharmacological preparation of Faecalibacterium prausnitzii strains. Preclinical murine study suggests that the administration of EXL01 could reverse the resistance to ICI induced by antibiotics (unpublished data).

We thus plan to test the concept of microbiota modification in patients treated with standard-of-care approved first-line immunotherapy for advanced HCC. We would include patients refractory to first-line treatment, and test the addition of EXL01 to standard-of-care approved first-line immunotherapy in order to reverse resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female
2. Age ≥18 years at time of signing informed consent
3. Presenting with HCC, diagnosed either by histological or radiological criteria as described by EASL
4. Locally advanced or metastatic and/or unresectable HCC according a Multidisciplinary Team meeting
5. Progressive disease after exposure to standard-of-care approved first-line immunotherapy
6. Decision made by the physician to continue the same standard-of-care approved first-line immunotherapy beyond progression
7. Child-Pugh A within 7 days prior to inclusion
8. ECOG performance status 0 to 1
9. Adequate hematological (Hemoglobin >8.5g/dL, platelets >60G/L, neutrophils >1.5G/L) and renal (creatinine clearance > 50 mL/min according to Cockcroft or MDRD formula) functions
10. Disease measurable by RECIST 1.1
11. Signed written Informed consent

Exclusion Criteria:

1. Partial response achieved under standard-of-care approved first-line immunotherapy
2. CTCAE Grade ≥3 or more toxicity under standard-of-care approved first-line immunotherapy, or persistent toxicity Grade >1
3. Liver involvement > 50%
4. Presence of major macro vascular invasion (except Vp1/Vp2)
5. Pregnant woman, or breastfeeding or women of child-bearing potential with no adequate contraception (see §4.3.1)
6. Under curatorship, guardianship, safeguard of justice or deprived of liberty
7. History of serious autoimmune disease
8. Interstitial lung disease
9. HBV chronic infection with HBV DNA > 100 IU/mL or without antiviral therapy; HBV patients with cirrhosis should be treated
10. HIV infection
11. Immunosuppression, including subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg/day prednisone equivalent)
12. Transplanted liver, or patient with intent for transplantation
13. Has difficulties in swallowing.
14. Has undergone major surgery or significant trauma ≤4 weeks prior to Screening. Note: Participants who had surgery >4 weeks prior to Screening must have recovered adequately from any toxicity and/or complications from the surgery or trauma prior to starting study intervention.
15. Is currently participating in or has participated in a study with an investigational compound or device within 3 months prior to the first dose of study intervention.

    Note: Participants who have entered the follow-up phase of an investigational study may participate so long as it has been at least 3 months since the last dose of the previous investigational agent.
16. Has a systemic infection or other serious infection requiring systemic treatment within 30 days prior to Screening.
17. Has a history of hypersensitivity to EXL01 and/or any excipients, which are listed in the IB, and/or to soybean or soy-containing products
18. Has a history of hypersensitivity to Chinese Hamster Ovary (CHO) cell products or other recombinant human or humanised antibodies
19. Active inflammatory intestinal disease (Crohn disease, Hemorrhagic recto-colitis, coeliac disease) or any serious chronic intestinal disease with uncontrolled diarrhea, or other inflammatory disease requiring anti-inflammatory medications
20. Current probiotics administration, or planned probiotics administration during treatment course.
21. Specific contra-indication to the continuation of the standard-of-care approved first-line immunotherapy :

21.1: for atezolizumab-bevacizumab:

* Thromboembolic events in the 3 months prior to inclusion
* Prior bleeding event due to untreated or incompletely treated esophageal and / or gastric varices within 6 months' prior inclusion
* Has a history of hypersensitivity to the atezolizumab or to any of the excipients listed in section 6.1 of the SmPC of atezolizumab
* Has a history of hypersensitivity to bevacizumab or to any of the excipients listed in section 6.1 of the SmPC of bevacizumab
* Uncontrolled hypertension
* Clinically significant cardiovascular disease such as pre-existing coronary artery disease, or congestive heart failure
* Proteinuria 21.2: for durvalumab:
* Has a history of hypersensitivity to the durvalumab or to any of the excipients listed in section 6.1 of the SmPC of durvalumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2026-03-12 (Estimated); Study Completion 2026-12-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate at week12 | At week12
  ORR defined as the best observed overall tumor response (BOR) from inclusion to W12, according RECIST 1.1 criteria
Adverse event | Maximum 15 month after le first EXL01 administration
  safety of atezolizumab-bevacizumab with bacterial supplementation EXL01

SECONDARY OUTCOMES:
Overall tumor response | At week6; at week12; at month 6, at month12
  Overall tumor response according to the mRECIST, RECIST 1.1 and iRECIST.
Objective Response Rate at week12 | at week 12
  ORR at week 12 according to mRECIST and iRECIST criteria
Objective Response Rate at M6 and M12 | At month 6, at month 12
  The ORR at M6, M12, according to the mRECIST, RECIST 1.1 and iRECIST criteria.
The Disease control rate (DCR), | At week12; at month 6, at month12
  The Disease control rate (DCR), as the proportion of patients with BOR as CR, PR or stable disease (SD) defined according to the mRECIST, RECIST 1.1 and iRECIST criteria at W12, M6, M12.
The Progression-Free Survival | Maximum 12 month after the fisrt EXL01 administration
  The Progression-Free Survival, defined as the time from patient inclusion to progression or death from any cause.
Overall survival (OS) | Maximum 15 month after the fisrt EXL01 administration of the last patient
  The Overall Survival, defined as the time from patient inclusion to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Héloise BOURIEN, Dr, Principal Investigator — Centre de lutte contre le cancer Eugène Marquis
Locations (6):
- France (6):
  - hôpital Avicenne, Bobigny
  - CHU de Bordeaux, Bordeaux
  - Hôpital Beaujon, Clichy
  - CHU de Nantes Hotel Dieu, Nantes
  - Centre de luttre contre le cancer Eugène Marquis, Rennes
  - Gustave ROUSSY, Villejuif

IPD SHARING:
Plan to Share IPD: No